CLINICAL TRIAL: NCT05935033
Title: A Phase 1, Open-label Trial to Evaluate the Pharmacokinetics and Safety Following a Single Dose of Emraclidine in Adult Participants With Mild, Moderate, and Severe Hepatic Impairment Compared With Adult Participants With Normal Hepatic Function
Brief Title: A Study to Evaluate the Effect of Hepatic Impairment on the Pharmacokinetics of Emraclidine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVL-231-SP-1008
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Hepatic Impairment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Severe Hepatic Impairment (Experimental): Participants will receive a single oral dose of 10 milligrams (mg) emraclidine.
  Interventions: Drug: Emraclidine
- Moderate Hepatic Impairment (Experimental): Participants will receive a single oral dose of 10 mg emraclidine.
  Interventions: Drug: Emraclidine
- Mild Hepatic Impairment (Experimental): Participants will receive a single oral dose of 10 mg emraclidine.
  Interventions: Drug: Emraclidine
- Normal Hepatic Function (Experimental): Participants will receive a single oral dose of 10 mg emraclidine.
  Interventions: Drug: Emraclidine

INTERVENTIONS:
Drug: Emraclidine — Tablet
  Other Names: CVL-231

SUMMARY:
The primary purpose of this study is to assess the effect of hepatic impairment on the pharmacokinetics (PK) of emraclidine following administration of a single oral dose in participants with mild, moderate, and severe hepatic impairment relative to matched participants with normal hepatic function.

ELIGIBILITY:
Key Inclusion Criteria:

1. All Participants

   - Male and female participants, body mass index of ≥18.0 to 42.0 kilograms per meter square (kg/m^2), inclusive, and a total body weight ≥50 kilograms (kg) (110 pounds [lbs]).
2. Additional Inclusion Criteria for Participants With Normal Hepatic Function

   * Participants who are healthy, having no clinically relevant abnormalities. Have normal hepatic function.
   * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), bilirubin and prothrombin time ≤ upper limit of normal (ULN) and albumin ≥ lower limit of normal (LLN) and ≤ ULN. Participants with a history of Gilbert syndrome are eligible provided direct bilirubin fraction is <20% of total bilirubin, and hemoglobin, and reticulocyte counts are all ≤ ULN.
3. Additional Inclusion Criteria for Participants With Hepatic Impairment - Participants with stable hepatic impairment that meets the criteria for Class A, Class B, or Class C of the modified Child-Pugh Classification. Stable hepatic disease defined as no clinically significant change in disease status in the last 28 days prior to the screening visit.

Key Exclusion Criteria:

1. For All Participants

   * Any condition or surgery that could possibly affect drug absorption, including, but not limited to, bowel resections, bariatric weight loss surgery/procedures, gastrectomy, and cholecystectomy.
   * Receipt of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccination or booster within 7 days of planned dosing.
   * Have recently been diagnosed with symptomatic coronavirus disease 2019 (COVID-19) or test positive for SARS-CoV-2 within 15 days prior to signing the informed consent form (ICF).
   * Positive drug screen or a positive test for alcohol at Screening or Baseline (Check-in/Day -1) Visits.
   * Use of prohibited medications prior to randomization or likely to require prohibited concomitant therapy during the trial.
   * Current use of tobacco or nicotine-containing products (cigarettes, cigars, chewing tobacco, snuff, e-cigarettes, etc). Note: Light smokers (<5 cigarettes/day or equivalent) are allowed provided they abstain from the use of tobacco- or nicotine-containing products for at least 2 hours prior to PK assessments.
   * Known allergy or hypersensitivity to the investigational medicinal product (IMP), closely related compounds, or any of their specified ingredients.
   * Has received IMP in a clinical trial of emraclidine within 12 months of signing the ICF.
   * Participants with a 12-lead ECG demonstrating any of the following at the Screening Visit and at Check-in (Day -1):

     * QT interval corrected for heart rate using Fridericia's formula (QTcF) interval >470 milliseconds (ms)
     * QRS interval >120 ms (unless right bundle branch block)
     * PR interval >200 ms
     * Left ventricular hypertrophy (LVH) with ST depressions and/or T wave inversions in leads with relatively tall R waves (ie, LVH with associated ST-T wave abnormalities)
     * Type 2 second-degree or third-degree atrioventricular block
     * Heart rate <45 beats per minute (bpm) or >100 bpm
     * Abnormal ECG changes (such as clinically significant ST depression or elevation or T wave inversion).
     * Abnormal heart rhythm (such as atrial fibrillation and atrial flutter)
   * Blood pressure measurements demonstrating any of the following at the Screening Visit and/or at Check-in (Day -1):

     * Supine systolic blood pressure ≥140 millimeters of mercury (mmHg) and/or diastolic blood pressure ≥90 mmHg
     * Standing systolic and/or diastolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg
     * Orthostatic hypotension, defined as a decrease of ≥20 mmHg in systolic blood pressure and/or ≥10 mmHg in diastolic blood pressure after at least 2 minutes of standing compared with the average of the resting supine blood pressure measurements.
2. Additional Exclusion Criteria for Participants with Hepatic Impairment

   * Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m^2 based on the Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) equation at Screening or Check-in (Day -1) visits
   * Acute hepatitis
   * Grade ≥2 hepatic encephalopathy
   * Participants who have received an organ transplant or are currently waiting for an organ transplant and are listed on the national transplant list.
   * Primary biliary cholangitis or primary sclerosing cholangitis
   * ALT or AST >5 × ULN or alkaline phosphatase >2 × ULN. Participants with a history of Gilbert syndrome are eligible provided direct bilirubin fraction is <20% of total bilirubin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Emraclidine | Pre-dose and at multiple timepoints post-dose up to Day 7
Maximum Observed Unbound Plasma Concentration (Cmax,u) of Emraclidine | Pre-dose and at multiple timepoints post-dose up to Day 7
Area Under the Plasma Concentration-time Curve from Time Zero to t (AUC0-t) of Emraclidine | Pre-dose and at multiple timepoints post-dose up to Day 7
Area Under the Unbound Plasma Concentration-time Curve from Time Zero to t (AUC0-t,u) of Emraclidine | Pre-dose and at multiple timepoints post-dose up to Day 7
Area Under the Plasma Concentration-time Curve from Time Zero to Infinity (AUCinf) of Emraclidine | Pre-dose and at multiple timepoints post-dose up to Day 7
Area Under the Unbound Plasma Concentration-time Curve From Time Zero to Infinity (AUCinf,u) of Emraclidine | Pre-dose and at multiple timepoints post-dose up to Day 7

SECONDARY OUTCOMES:
Incidence and Severity of Treatment Emergent Adverse Events (TEAEs) | Day 1 up to Follow-up (Day 15)
Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Values | Days 1 to 7
Number of Participants With Clinically Significant Changes in Vital Signs | Days 1 to 7
Number of Participants With Clinically Significant Changes in Laboratory Assessments | Days 1 to 7
Number of Participants With Clinically Significant Changes in Physical and Neurological Examination Results | Days 1 to 7
Changes in Columbia Suicide Severity Rating Scale (C-SSRS) Score | Days 1 to 7
  The C-SSRS includes 'yes' or 'no' responses for assessment of suicidal ideation and behavior as well as numeric ratings for severity of ideation, if present (from 1 to 5, with 5 being the most severe). Greater lethality or potential lethality of suicidal behaviors (endorsed on the behavior subscale) indicates increased risk.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (3):
- United States (3):
  - Miami, Florida, Miami, Florida
  - Orlando, Florida, Orlando, Florida
  - San Antonio, Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No